CLINICAL TRIAL: NCT01289665
Title: The Effect of Lubricating Gel on Patient Comfort During Speculum Insertion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Principal Investigator, D. Ashley Hill, MD, Associate Director, Department of Obstetrics and Gynecology, AdventHealth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2644-7780
Record Dates: First submitted 2011-02-02; First posted 2011-02-04 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Examination, Gynecological; Examination, Pelvic; Examination, Vaginal
Keywords: lubricating; gel; speculum; Pain, Pelvic; Examination, Gynecological
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubricating Gel (Experimental)
  Interventions: Procedure: Lubricating gel used during speculum insertion.
- Water (Active Comparator)
  Interventions: Procedure: Water used during speculum examination.

INTERVENTIONS:
Procedure: Lubricating gel used during speculum insertion. — Examiner will use 0.5 mL of sterile lubricating gel to lubricate standard-sized plastic speculum during clinically indicated vaginal speculum examination. Patients will mark visual analog scale immediately following insertion.
  Arms: Lubricating Gel
Procedure: Water used during speculum examination. — Patients will under vaginal speculum examination using 3 mL of water as a lubricant and will mark a visual analog scale immediately after speculum insertion.
  Arms: Water

SUMMARY:
The purpose of this study is to determine if lubricating gel affects patients' perception of discomfort during speculum insertion, as compared to water.

DETAILED DESCRIPTION:
The outcome measure is patient discomfort as measured by a visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing vaginal speculum examination between the ages of 18 and 50.

Exclusion Criteria:

* Pregnancy.
* Non-English speaking.
* Using hormone therapy.
* Active vulvar or vaginal lesion, infection or complaint.
* Undergoing vaginal or vulvar procedure or biopsy.
* History of chronic pelvic pain, interstitial cystitis or vulvar vestibulitis.
* History of prior vulvar or vaginal surgical procedures.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Hill, MD, Study Chair — AdventHealth
Locations (1):
- Department of Obstetrics and Gynecology, Florida Hospital, Orlando, Florida, United States

REFERENCES:
- [Derived] Hill DA, Lamvu G. Effect of lubricating gel on patient comfort during vaginal speculum examination: a randomized controlled trial. Obstet Gynecol. 2012 Feb;119(2 Pt 1):227-31. doi: 10.1097/AOG.0b013e3182426275. PMID 22270273

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lubricating Gel | Water
Started | 60 | 60
Completed | 59 | 60
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubricating Gel | Water | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 60 | 119
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 60 | 119
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 55 | 54 | 109
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient Discomfort During Speculum Insertion as Measured by a Visual Analog Scale.
Description: The outcome measure is a single measurement of pain using a 10-point visual analog scale entitled "Visual Pain Scale" immediately following speculum insertion. The scale is a continuous 10cm line with the minimum value of 0 (labeled "no pain") on the left side of the line, and a maximum value of 10 (labeled "worst pain") on the right side of the line. Higher scores represent more pain and a worse outcome. There are no additional measurements obtained, and patients will not be followed for study purposes thereafter.
Time Frame: Immediate.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubricating Gel | Water
Number analyzed (Participants) | 59 | 60
score on a scale | 1.41 (1.55) | 2.15 (1.93)

ADVERSE EVENTS:
Arm/Group | Lubricating Gel | Water
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 0/59 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes